CLINICAL TRIAL: NCT07217431
Title: Access BNP on DxI 9000 Clinical Performance Evaluation: Specimen Testing and Clinical Concordance Study
Brief Title: Access BNP Clinical Performance Evaluation: Testing and Clinical Concordance Study
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BNP-02-23
Record Dates: First submitted 2025-06-03; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects with heart failure: Targeting subjects in the acute care setting that present with suspicion of either new onset or worsening symptoms of heart failure
  Interventions: Diagnostic Test: BNP

INTERVENTIONS:
Diagnostic Test: BNP — Blood collected during this study will be tested on separate IUO BNP assay on a separate protocol. No active interventions will occur during this study.

SUMMARY:
The goal is to establish clinical performance of a BNP assay on the intended use population and establish clinical concordance on a separate device.

ELIGIBILITY:
Inclusion Criteria:

* There is no direct inclusion criteria for this study, Samples were collected under a separate enrollment protocol

Exclusion Criteria:

* Hemolysis observed per CLSIC56A grading scale
* Icterus (bilirubin) observed 4+ per CLSIC56A grading scale

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specimens are to be collected under BNP-05-24 protocol are used. Approximately 1100 K2 EDTA samples with concentrations that span the analytical measuring range (AMR) are used in this testing study.
Sampling Method: Non-Probability Sample
Enrollment: 1361 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Heart failure positive subjects | Through study completion, approximately 9 months
  Subjects with BNP value above clinical decision point

SECONDARY OUTCOMES:
Heart failure negative subjects | Through study completion, approximately 9 months
  Subjects with BNP value below clinical decision point

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Maryland-Baltimore, Baltimore, Maryland
  - HealthPartners Central Laboratory, Eden Prairie, Minnesota
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT07217431/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT07217431/SAP_001.pdf